CLINICAL TRIAL: NCT01102491
Title: The Effect of Multimodal Anti-emetic Protocol on Postoperative Nausea and Vomiting After Total Knee Arthroplasty
Brief Title: Additional Anti-emetic Effect of Ramosetron Prophylaxis After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B-1001/091-003
Record Dates: First submitted 2010-04-08; First posted 2010-04-13 (Estimated); Results first posted 2010-05-21 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Osteoarthritis, Knee
Keywords: postoperative nausea and vomiting
MeSH Terms: conditions — Osteoarthritis, Knee; Postoperative Nausea and Vomiting | interventions — ramosetron

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ramosetron prophylaxis (Experimental): ramosetron prophylaxis at the end of surgery with starting PCA and 1 day after surgery
  Interventions: Drug: Ramosetron
- Control (No Intervention): no antiemetic prophylaxis

INTERVENTIONS:
Drug: Ramosetron — ramosetron intravenous injection, 0.3mg, 1 time/day for 2 days
  Other Names: Nasea
  Arms: Ramosetron prophylaxis

SUMMARY:
The purposes of this study are to document the antiemetic efficacy of multimodal antiemetic protocol in patient after Total Knee Arthroplasty using regional anesthesia, midazolam & propofol, hydration & oxygen supplement, preemptive & multimodal contemporary pain management and to determine whether Ramosetron prophylaxis would provide additional antiemetic effect on this protocol. We hypothesized that the incidence of Postoperative nausea and vomiting during multimodal antiemetic protocol would be lower than Apfel's expected postoperative nausea and vomiting incidence. It was also hypothesized that Ramosetron prophylaxis would provide additional antiemetic effect.

DETAILED DESCRIPTION:
Immediate postoperative pain after Total Knee Arthroplasty(TKA) remains an unsolved problem, and a substantial proportion of patients experience moderate to severe postoperative pain. Patient controlled analgesia(PCA) using opioid is an effective and safe modality for postoperative pain relief after TKA and remains an integral part of pain management after TKA. However, Opioid is associated with high incidence of postoperative nausea and vomiting(PONV) which is the most frequent complication during the first 24 hour after surgery.PONV has been reported to be more distressing than postoperative pain and to be the most undesirable negative outcome. Despite advances in prevention and treatment of PONV, PONV remains a continuing problem with an incidence of 20-30% in unselected patients and up to 70% in "high-risk" patients. As results of current researches, some risk factors of PONV have been identified and indications of prophylactic antiemetics and strategies to reduce baseline risk have been recommended.The recommended modalities to reduce baseline risk includes regional anesthesia, oxygen supplement, use of midazolam and propofol and avoid use of inhaled anesthesia and neuromuscular blockade. In addition,published evidence suggests that appropriate antiemetic prophylaxis should be considered for patients with 2 or more risk factors and to reduce opioid consumption, preemptive multimodal pain management such as preemptive analgesic medication, continuous regional nerve block is recommended.Ramosetron is a newly developed serotonin receptor antagonist with a higher affinity and longer duration of action than that of the previously developed serotonin receptor antagonist such as ondansetron and granisetron. Thus, this prospective blinded randomized study was conducted to document the antiemetic efficacy of multimodal antiemetic protocol to reduce baseline risk, using regional anesthesia, midazolam and propofol, hydration and oxygen supplement and multimodal pain control protocols using the continuous femoral nerve block, PCA and preemptive oral medications and to determine whether Ramosetron prophylaxis would provide additional antiemetic effect in patients after TKA for whom covered by this multimodal antiemetic protocols.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary osteoarthritis, knee
* Scheduled for elective total knee arthroplasty
* Signed written informed consent

Exclusion Criteria:

* Refusing participate
* Contraindication to regional anesthesia
* Severe impairment of bowel motility
* administration of other antiemetics within 24hours before surgery
* systemic steroid within 24hours before surgery
* history of cardiovascular & respiratory disease
* renal & hepatic failure

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T K Kim, MD,PhD, Principal Investigator — Joint Recontruction Center, Seoul National University Bundang hospital
Locations (1):
- Joint Reconstruction Center, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 153 patients whose diagnosis was primary osteoarthritis scheduled for unilateral total knee arthroplasty(TKA)at Seoul National University Bundang Hospital from October 2009 to March 2010 were recruited.
Pre-assignment Details: 11 patients were excluded before assignment. 6 were other diagnosis such as rheumatoid arthritis, secondary osteoarthritis, 2 were refused to participate this study, and 3 were serious medical conditions such as respiratory failure, heart failure.
Period: Overall Study
Arm/Group | Ramosetron Prophylaxis | Control
Started | 71 | 71
Completed | 60 (11 patient excluded) | 59 (12 patients were excluded)
Not Completed | 11 | 12
Not completed — Protocol Violation | 11 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramosetron Prophylaxis | Control | Total
Number analyzed (Participants) | 71 | 71 | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 16 | 29
  >=65 years | 58 | 55 | 113
Age Continuous [Mean (Standard Deviation); unit: years] | 69.1 (6.3) | 69.0 (7.5) | 69.1 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 65 | 129
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 71 | 71 | 142

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Nausea and Vomiting
Description: outcomes assessor who is blinded to randomization assessed the incidence of postoperative nausea which was defined as subjectively unpleasant sensation associated with awareness of the urge to vomit and an emetic episode and vomiting
Time Frame: within 48 hours after surgery
Measure: Number; unit: participants
Arm/Group | Ramosetron Prophylaxis | Control
Number analyzed (Participants) | 71 | 71
participants | 25 | 32
Statistical Analysis 1: Comparison: Ramosetron Prophylaxis vs Control; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Incidence of Rescue Antiemetic Administration
Description: outcome assessor assessed the incidence of rescue antiemetic administration
Time Frame: within 48 hours after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Ramosetron Prophylaxis | Control
Serious Adverse Events (participants affected / at risk) | 27/71 | 25/71
Other Adverse Events (participants affected / at risk) | 4/71 | 2/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ramosetron Prophylaxis (N=71) | Control (N=71)
Drowsiness (Nervous system disorders) | 27 | 25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ramosetron Prophylaxis (N=71) | Control (N=71)
headache (Nervous system disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No